CLINICAL TRIAL: NCT06128083
Title: Prelimenary Observational Study of the Influence of Adherence to the Recommandations Issued by the National Nutrition and Health Program on the Risk of Overweiht and Obesity in Children : the Case of a Municipality That Has Signed the " Ville Active PNNS " Charter
Brief Title: Evaluation of the Impact of Eating Habits on Children's Corpulence
Acronym: KALI SANTE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22-PP-05
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood
Keywords: Child; Obesity; Alimentation; Nutrition
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Childhood obesity has been rising steadily over the past 40 years. In 2016, the World Health Organization (WHO) observed around 340 million overweight or obese children and adolescents worldwide, including one in five in France. The causes are complex, both individual (genetic, biological, behavioral) and collective (social, economic, cultural). Childhood obesity encourages the development of chronic diseases such as diabetes and hypertension, and can affect mental health. Without early treatment, the risk of obesity persisting into adulthood is high.

In the Alpes-Maritimes region, the commune of Mouans-Sartoux has been promoting a local diet in line with PNNS-4 recommendations since 2011.

We wish to study the impact of these actions on the health of Mouans children. We propose a preliminary observational study to assess the relationship between family adherence to PNNS recommendations and the prevalence of overweight and obesity in Mouans-Sartoux elementary school children.

ELIGIBILITY:
Inclusion Criteria:

* The child must be enrolled in one of Mouans-Sartoux's three public elementary school (A. Legall / F. Jacob / Orée du bois) at the start of the 2023 school year
* Social Security affiliation
* Non-opposition of the legal representative(s) of parental authority

Exclusion Criteria:

* Opposition to participation in research involving the human person
* In the event of disagreement between the parents, we will take non-participation into account

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children enrolled in one of Mouans-Sartoux's 3 public elementary school.
  * Schools (3): A. Legall / F. Jacob / Orée du bois.
  * Classes: CP to CM2 inclusive.
  * There are no age or gender restrictions. Children not enrolled in the school canteen may participate.
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
To assess the association between the risk of overweight and/or obesity in children and family adherence to PNNS-4 recommendations. | 1 year
  Calculation of the odd-ratio (OR) between the risk of "overweight and/or obesity" in children (corresponding to a BMI z-score > 1) and family adherence to PNNS recommendations estimated from the "PNNS-GS2" score using a univariate logistic regression model.

SECONDARY OUTCOMES:
To assess the association between the risk of overweight and/or obesity in children and the importance of organic food in family dietary habits. | 1 year
  The "Organic and Local Food Consumption" questionnaire (18) is used to estimate household consumption of organic products. The score obtained from this questionnaire will be evaluated in a similar way to the "PNNS-GS2" score.
  We will study the prevalence of overweight and obesity according to the presence or absence of each listed risk factor belonging to the following categories:
  * Children's physical activity and sports
  * Favorable behaviors
  * Household socio-demographic data
  * Child's environment
  * Parents' lifestyle
  * Declarative medical data
Evaluate the influence of children's school canteen enrolment on family adherence to the National Health Nutrition Program 4 (PNNS-4) recommendations by PNNS-GS2) score | 1 year
  We will assess the impact of whether or not children are enrolled in the canteen by studying for each group the distribution of the National Health Nutrition Program - Guidelines Score 2 (PNNS-GS2) score; The "PNNS-GS2" score assesses families' adherence to the PNNS-4 recommendations, based on a list of items relating to eating habits. Responses are grouped into quartiles to form comparison groups. In this study, the score is assessed at family level.
Evaluate the influence of children's school canteen enrolment on family adherence to the National Health Nutrition Program 4 (PNNS-4) recommendations by "Organic and Local Food Consumption" score | 1 year
  We will assess the impact of whether or not children are enrolled in the canteen by studying for each group the distribution of the "Organic and Local Food Consumption" score.
  List of food groups
  1. Fruit
  2. Vegetables
  3. Soy
  4. Dairy products
  5. Meat and fish
  6. Eggs
  7. Grains and pulses
  8. Bread and cereals
  9. Flour
  10. Vegetable oils and condiments
  11. Prepared dishes
  12. Coffee/tea/tea tea
  13. Sweet products
  14. Food supplements
  15. Other foods
  For each group, participants indicated their frequency of consumption
  * Organic: "Most of the time", "From time to time", "Never".
  * Locally produced: "Most of the time", "From time to time", "Never".
  Two scores are created: "organic food score" for organically sourced food, and "local food score" for locally produced food, awarding:
  * 2 points for "Most of the time
  * 1 point for "Once in a while
  * 0 points for "Never The two scores are added together to obtain the "organic and local food score".
Evaluate the influence of children's school canteen enrolment on family adherence to the National Health Nutrition Program 4 (PNNS-4) recommendations by the distribution of the z-score. | 1 year
  We will assess the impact of whether or not children are enrolled in the canteen by studying for each group the distribution of the z-score and the prevalence of overweight and obesity.
  In children, BMI is not a good representation of corpulence, as individual growth varies according to sex and age. We therefore use the BMI z-score (called "Z-score" in this study), which expresses the deviation of a child's BMI from the reference value according to sex and age.
  The Z-score can be used to classify children into several categories according to the following limits:
  * Extreme thinness
  * Thin
  * Normal build
  * Overweight
  * Obese
Evaluate the influence of children's school canteen enrolment on family adherence to the National Health Nutrition Program 4 (PNNS-4) recommendations by prevalence of risks factors. | 1 year
  We will assess the impact of whether or not children are enrolled in the canteen by studying for each group prevalence of risk factors studied.
Compare the observed proportion of mouansois children who are overweight or obese with data from the Alpes-Maritimes department's maternal and child protection service. | 1 year
  We will calculate the difference between the observed proportion of overweight or obese children in Mouans and that expected according to the data presented by the Protection Maternelle et Infantile des Alpes-Maritimes.
Collect hair samples from local children to build up a sample bank for future research into the presence of pesticides and endocrine disruptors. | 1 year
  We will be collecting hair samples from volunteer children in Mouans, in order to build up a sample bank in parallel with the study, with a view to future work on measuring the presence of endocrine disruptors / pesticides.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin LEGUEULT, MD, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice - Hôpital Archet 1, Nice, Alpes-Maritimes, France